CLINICAL TRIAL: NCT03010644
Title: Summer Weight and Environmental Assessment Trial (SWEAT)
Brief Title: Summer Weight and Environmental Assessment Trial
Acronym: SWEAT
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: USDA North Central - Nutrition Education Center of Excellence (Unknown)
Responsible Party: Principal Investigator, Carolyn Gunther, Assistant Professor, Ohio State University
Other Study IDs: 2016B0034
Record Dates: First submitted 2016-12-21; First posted 2017-01-05 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2017-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Underserved school-aged children: Underserved school-aged children at risk for obesity
  Interventions: Other: n/a - observational study

INTERVENTIONS:
Other: n/a - observational study — n/a - observational study

SUMMARY:
The consequences of childhood obesity are devastating, affecting the physical and mental health of children. Disadvantaged school-age children are at risk for unhealthy gains in BMI during the summer months and there is a dearth of information regarding the causal health behaviors and environmental factors. The overall objective of this application is to provide an in depth examination of key dietary and physical activity behaviors as well as the food, physical activity, and social environments of low-income, racial/ethnic school-age children. To achieve this goal, an observational study utilizing a multi-state prospective cohort design will be conducted with the goal of examining the weight gain trajectory among a racially and ethnically diverse convenience sample of disadvantaged school-age children who routinely attend structured programming during the summer months and those who don't participate in structured programming. In addition, a subset of these children will be evaluated to learn their daily health behaviors, as well as their food, physical activity, and social environments during the summer. Identification of determinants of program participation and factors that may enhance the beneficial effects of program participation will also occur. A social ecological framework approach will guide the research. This study can be expected to have a significant positive impact by providing information on the factors that protect disadvantaged children from unhealthy weight gain during the summer which can be used by stakeholders at the local, state, and federal level to reform current policy that will increase child participation in health promoting programming during the summer window of risk.

ELIGIBILITY:
Inclusion Criteria:

* School-aged children (rising kindergartners through rising 5th graders) attending schools in the target neighborhoods.

Exclusion Criteria:

* None

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Racially and ethnically diverse convenience sample of disadvantaged school-age children
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in BMI | Baseline (beginning of summer), T1 (5 weeks), T2 (10 weeks), T3 (22 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Purdue University, West Lafayette, Indiana
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hopkins LC, Tiba S, Westrick M, Gunther C. The Diet Quality of a Sample of Predominantly Racial Minority Children From Low-Income Households Is Lower During the Summer vs School Year: Results From the Project Summer Weight and Environmental Assessment Trial Substudy. J Acad Nutr Diet. 2021 Jan;121(1):112-120. doi: 10.1016/j.jand.2020.06.013. Epub 2020 Aug 14. PMID 32800759
- [Derived] Hopkins LC, Penicka C, Evich C, Jones B, Gunther C. Project SWEAT (Summer Weight and Environmental Assessment Trial): study protocol of an observational study using a multistate, prospective design that examines the weight gain trajectory among a racially and ethnically diverse convenience sample of economically disadvantaged school-age children. BMJ Open. 2018 Aug 29;8(8):e021168. doi: 10.1136/bmjopen-2017-021168. PMID 30158223